CLINICAL TRIAL: NCT03296410
Title: The Safety and Immunogenicity of Enterovirus Type 71 Inactivated Vaccine (Human Diploid Cell) With Two Measles Attenuated Live Vaccine and Live Attenuated Japanese Encephalitis Vaccine at the Same Time Point in Infants (8-month-old)
Brief Title: The Phase IVd of Inactivated Enterovirus 71 Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Guangdong Center for Disease Prevention and Control (Other Government)
Responsible Party: Principal Investigator, Qihan Li, Professor, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20170710
Record Dates: First submitted 2017-09-01; First posted 2017-09-28 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Hand, Foot and Mouth Disease (HFMD)
Keywords: Hand, Foot and Mouth Disease (HFMD); immunogenicity; safety
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- EV71 and two measles attenuated live vaccine (Experimental): infants vaccinated with enterovirus type 71 inactivated vaccine (human diploid cell) and two measles attenuated live vaccine at 8 months old, and vaccinated with the second dose of enterovirus type 71 inactivated vaccine (human diploid cell) at 9 months old.
  Interventions: Biological: EV71 and two measles attenuated live vaccine
- EV71 and attenuated Japanese encephalitis vaccine (Experimental): infants vaccinated with enterovirus type 71 inactivated vaccine (human diploid cell) and live attenuated Japanese encephalitis vaccine at 8 months old, and vaccinated with the second dose of enterovirus type 71 inactivated vaccine (human diploid cell) at 9 months old.
  Interventions: Biological: EV71 and attenuated Japanese encephalitis vaccine
- two measles attenuated live vaccine (Active Comparator): infants vaccinated with two measles attenuated live vaccine at 8 months old
  Interventions: Biological: two measles attenuated live vaccine
- live attenuated Japanese encephalitis vaccine (Active Comparator): infants vaccinated with live attenuated Japanese encephalitis vaccine at 8 months old
  Interventions: Biological: live attenuated Japanese encephalitis vaccine
- EV71 vaccine (Active Comparator): infants vaccinated with enterovirus type 71 inactivated vaccine (human diploid cell) at 8 months old, and vaccinated with the second dose of enterovirus type 71 inactivated vaccine (human diploid cell) at 9 months old.
  Interventions: Biological: EV71 vaccine

INTERVENTIONS:
Biological: EV71 and two measles attenuated live vaccine — infants vaccined with two dose (3.0 EU/dose) of inactivated enterovirus 71 vaccine (KMB-17) at 8 months old and 9 months old (namely interval one month). And meanwhile, they routine vaccined with two measles attenuated live vaccine at 8 months old.
  Arms: EV71 and two measles attenuated live vaccine
Biological: EV71 and attenuated Japanese encephalitis vaccine — infants vaccined with two dose (3.0 EU/dose) of inactivated enterovirus 71 vaccine (KMB-17) at 8 months old and 9 months old (namely interval one month). And meanwhile, they routine vaccined with attenuated Japanese encephalitis vaccine at 8 months old.
  Arms: EV71 and attenuated Japanese encephalitis vaccine
Biological: two measles attenuated live vaccine — infants vaccined with one dose two measles attenuated live vaccine at 8 months old.
  Arms: two measles attenuated live vaccine
Biological: live attenuated Japanese encephalitis vaccine — infants vaccined with one dose attenuated Japanese encephalitis vaccine at 8 months old.
  Arms: live attenuated Japanese encephalitis vaccine
Biological: EV71 vaccine — infants vaccined with two dose (3.0 EU/dose) of inactivated enterovirus 71 vaccine (KMB-17) at 8 months old and 9 months old (namely interval one month).
  Arms: EV71 vaccine

SUMMARY:
Enterovirus 71 (EV71), a major pathogen causing hand-foot-and-mouth disease (HFMD) worldwide, is a member of the Human Enterovirus species A, family Picornaviridae. Its infection occasionally leads to severe diseases and death, with central nervous system (CNS) damage.

Recently, except of inactivated vaccine, several EV71 vaccine candidates have been evaluated in animals but no final results of clinical trials, such as attenuated vaccine, subunit vaccine. A formalin-inactivated EV71 vaccine (Human Diploid cell, KMB-17 Cell) has been finished phase I, II and III clinical trials and licensed by SFDA in China at Dec. 3, 2015. Based on the results of clinical trials, the protective efficacy of inactivated EV71 vaccine is 97% against HFMD caused by EV71. The phase IV clinical trial has been carried out from July 2016. The purpose of phase IVd is to evaluated the immunogenicity and safety of the inactive EV71 vaccine within two measles attenuated live vaccine and live attenuated Japanese encephalitis vaccine at the same time point in large scale population of Chinese children (8 months old) in Guangdong Province, China.

DETAILED DESCRIPTION:
There are two parts of phase IVd clinical trials have been performed. First, to evaluate the immunogenicity of the inactive EV71 vaccine within two measles attenuated live vaccine and live attenuated Japanese encephalitis vaccine at the same time point in large scale population of Chinese children (8 months old), within 56-day-post-immunized.

Second, to safety of the inactive EV71 vaccine within two measles attenuated live vaccine and live attenuated Japanese encephalitis vaccine at the same time point in large scale population of Chinese children (8 months old), within 56-day-post-immunized.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects (6-71 months old children) as established by medical history and clinical examination
* The subjects' legal guardian must be aware of this vaccines
* The subjects' legal guardian voluntarily participate in the study and signed Informed Consent Form
* Subjects with temperature ≤ 37.0 ℃
* The subjects' legal guardian with the ability and objective to comply with the requirements of the protocol
* Persist for a 14-month visit (and receive blood, stool (or specimens by means of a swab) tests according to program requirements in immunogenicity observation group)

Exclusion Criteria:

* Allergy or serious side-effects to a vaccine or any ingredient of vaccine
* Epilepsy, seizures, convulsions, neurological illness
* Congenital or hereditary immunodeficiency
* Autoimmune disease
* Asthma, thyroidectomy, angioneurotic edema, diabetes or cancer
* Asplenia, functional asplenia, and any circumstances leading to the asplenia or splenectomy
* Clinical diagnosis of coagulopathy (such as clotting factor deficiency, coagulation disorders, platelet abnormalities), significant bruising or blood clotting disorder
* Acute illness or acute exacerbation of chronic disease in last 7 days
* Any prior administration of immunodepressant or corticosteroids in last 6 months
* Any prior administration of blood products in last 3 months
* Any prior administration of live-attenuated vaccine in last 15 days
* Any prior administration of subunit or inactivated vaccines in last 7 days
* Fever before vaccination, axillary temperature ﹥37.0 ℃
* The laboratory test abnormalities before vaccination, including blood tests (hemoglobin, total white blood cells, WBC, platelets), blood biochemistry tests (ALT, total bilirubin, direct bilirubin, Cr, BUN) and urine tests (urine protein, urine sugar, blood cells), etc.
* Hypertension or hypotension. Systolic blood pressure ﹥140 mmHg and/ or diastolic blood pressure ﹥90 mmHg; systolic blood pressure ﹤90 mmHg and/or diastolic blood pressure ﹤60 mmHg
* Any condition that in the opinion of the investigator, may interfere with the evaluation of study objectives
* take part into other vaccine or drug clinical trials in last half year

Ages: 8 Months to 9 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1220 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-09-02 (Estimated); Study Completion 2019-09-02 (Estimated)

PRIMARY OUTCOMES:
Evaluate the seropositive rate of anti-EV71 antibodies in serum of children before first vaccination | at 0 day before finishing 1st doses immunization
  Bloods were obtained before first vaccination. The antibody titers were tested in serum of children.
Evaluate the seropositive rate of anti-EBV antibodies in serum of children before first vaccination | at 0 day before finishing 1st doses immunization
  Bloods were obtained before first vaccination. The antibody titers were tested in serum of children.
Evaluate the seropositive rate of anti-measles virus antibodies in serum of children before first vaccination | at 0 day before finishing 1st doses immunization
  Bloods were obtained before first vaccination. The antibody titers were tested in serum of children.
Evaluate the seropositive rate of anti-Rubella virus antibodies in serum of children before first vaccination | at 0 day before finishing 1st doses immunization
  Bloods were obtained before first vaccination. The antibody titers were tested in serum of children.
Evaluate the seroconversion rate of anti-EV71 antibodies in serum of children at 56 days after first vaccination | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children.
Evaluate the seroconversion rate of anti-EBV antibodies in serum of children at 56 days after first vaccination | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children.
Evaluate the seroconversion rate of anti-measles virus antibodies in serum of children at 56 days after first vaccination | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children.
Evaluate the seroconversion rate of anti-Rubella virus antibodies in serum of children at 56 days after first vaccination | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children.

SECONDARY OUTCOMES:
Evaluate the antibody titers of anti-EV71 antibodies in serum of children | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children at 56 days.
Evaluate the antibody titers of anti-EBV antibodies in serum of children | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children at 56 days.
Evaluate the antibody titers of anti-measles virus antibodies in serum of children | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children at 56 days.
Evaluate the antibody titers of anti-Rubella virus antibodies in serum of children | at 56 days after finishing 1st doses immunization
  Bloods were obtained at 56 days after first vaccination. The antibody titers were tested in serum of children at 56 days.
Incidence of treatment adverse events finishing 1st doses immunization | within 28 days after finishing 1st doses immunization
  The adverse events were observed and recorded within 30 minutes post immunization (p.i.), within 0-1 days post immunization (d.p.i.), within 1-3 d.p.i. and within 28 d.p.i. after the 1st injection.
Incidence of treatment adverse events finishing 2nd doses immunization | within 28 days after finishing 2nd doses immunization
  The adverse events were observed and recorded within 30 minutes post immunization (p.i.), within 0-1 days post immunization (d.p.i.), within 1-3 d.p.i. and within 28 d.p.i. after injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Province Center for Diseases Control and Prevention, Guangzhou, Guangdong, China